CLINICAL TRIAL: NCT04569643
Title: Periodic Limb Movement Syndrome in Patients With Cerebral Small Vessel Disease: a Clinical and Neuropsychological Study.
Brief Title: Periodic Limb Movement Syndrome in Patients With Cerebral Small Vessel Disease.
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 2207
Record Dates: First submitted 2020-09-24; First posted 2020-09-30 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2020-08

CONDITIONS: Periodic Limb Movement Disorder; Cerebral Small Vessel Diseases; Cognitive Dysfunction
Keywords: Aged; Cerebral Small Vessel Disease; Cognitive Dysfunction; Magnetic Resonance Imaging; Periodic Limb Movement Disorder; Sleep Disorder
MeSH Terms: conditions — Nocturnal Myoclonus Syndrome; Cerebral Small Vessel Diseases; Cognitive Dysfunction; Sleep Wake Disorders | interventions — Actigraphy; Neuroimaging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Main: Patients with cerebral small vessel disease and periodic limb movement index equal or more than 15 movements per hour of sleep.
  Interventions: Diagnostic Test: Actigraphy; Diagnostic Test: Cardiorespiratory monitoring; Diagnostic Test: Neuroimaging; Other: Assessment of cognitive function; Other: Sleep quality and mood questionnaires
- Control: Patients with cerebral small vessel disease and periodic limb movement index less than 15 movements per hour of sleep.
  Interventions: Diagnostic Test: Actigraphy; Diagnostic Test: Cardiorespiratory monitoring; Diagnostic Test: Neuroimaging; Other: Assessment of cognitive function; Other: Sleep quality and mood questionnaires

INTERVENTIONS:
Diagnostic Test: Actigraphy — Participants will undergo overnight leg actigraphy at baseline. Leg movements will be recorded bilaterally by actigraphic method with two ankle-worn recorders.
Diagnostic Test: Cardiorespiratory monitoring — All participants will be scanned for presence of sleep-related breathing disorders with a portable monitoring device at baseline. The compact screening device will be attached to the patient's wrist during the night sleep.
Diagnostic Test: Neuroimaging — All subjects will undergo brain MRI scanning at baseline and in 1-year follow-up. The imaging protocol will include axial T1, T2, T2*, FLAIR and diffusion-weighted imaging scans that will be made on a 3-Tesla scanner.
Other: Assessment of cognitive function — Assessment will take place at weeks 0 (baseline) and 52 (1 year follow-up). The neuropsychological protocol will be consist of Montreal Cognitive Assessment (MoCA), 12-word Verbal Memory Test, Benton Visual Retention Test, Frontal Assessment Battery, Trail Making Test (parts A and B), phonetic (as a part of the MoCA) and semantic verbal fluency assessment, Symbol Digit Modalities Test.
Other: Sleep quality and mood questionnaires — Self-reporting scales and questionnaires will be used at baseline to assess sleep quality, daytime functioning and mood. The protocol includes the Pittsburgh Sleep Quality Index, the Epworth Sleepiness Scale, the Geriatric Depression Scale.

SUMMARY:
Patients from 60 to 75 years old diagnosed with cerebral small vessel disease with no history of symptomatic stroke, brain tumor, traumatic brain injury, seizures and neurodegenerative or mental disorder will undergo overnight leg actigraphy and cardiorespiratory monitoring. Those of them with apnea/hypopnea index under 5 will be enrolled. Brain MRI and cognitive assessment will be performed at baseline and in 1-year follow-up, sleep quality will be assessed at baseline with self-reported questionnaires. Progression of cerebral small vessel disease markers and cognitive dysfunction will be compared between patients with high periodic limb movement index (the number of periodic limb movement ≥ 15 per hour of sleep) and controls (periodic limb movement index < 15/h).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a cerebral small vessel disease - assessed by MRI.
* Ability to follow the procedures of the study, fluent Russian language - assessed by self-report.

Exclusion Criteria:

* History of symptomatic stroke, brain tumor or traumatic brain injury - assessed by self-report and clinical history.
* History of severe psychiatric comorbidities other than anxiety and depression, substance use disorder - assessed by self-report and clinical history.
* Significant visual loss (leading to difficulties with performing cognitive tasks) - assessed by self-report and clinical history.
* Presence of dementia - assessed by history and clinical examination.
* Movement disorders (e.g. tremor, dystonia etc.) leading to lower velocity of performing cognitive tasks against the clock - assessed by clinical examination.
* Obstructive sleep apnea syndrome - according to the criteria of International classification of sleep disorders III.
* Restless legs syndrome - according to the criteria of the International restless legs syndrome study group.
* Current intake of neuroleptics, benzodiazepines, selective serotonin reuptake inhibitors - assessed by self-report and clinical history.

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with сerebral small vessel disease will be recruited among in-hospital patients (1st and 2nd Department of Neurology, University clinic 3, Sechenov First Moscow State Medical University, Moscow).
Sampling Method: Probability Sample
Enrollment: 76 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
White matter hyperintensities volume change | 1 year
  All the images will be processed with online software pipeline to make an automated volumetric measurement of white matter hyperintensities. The volume of the white matter lesion will be calculated separately for the periventricular, juxtacortical, infratentorial and deep white matter areas as well as total volume of the lesion. Baseline volumes will be subtracted from follow-up volumes to obtain absolute white matter hyperintensities volume change.
Degree of Cognitive Decline | 1 year
  The scores of cognitive tests (Montreal Cognitive Assessment (MoCA), 12-word Verbal Memory Test, Benton Visual Retention Test, Frontal Assessment Battery, Trail Making Test (parts A and B), phonetic and semantic verbal fluency assessment, Symbol Digit Modalities Test) at baseline will be subtracted from the corresponding baseline scores. The obtained difference reflects the degree of cognitive decline in 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Ekaterina D. Spektor, M.D., Principal Investigator — I.M. Sechenov First Moscow State Medical University (Sechenov University)
Locations (1):
- I.M. Sechenov First Moscow State Medical University (Sechenov University), Moscow, Russia

IPD SHARING:
Plan to Share IPD: No